CLINICAL TRIAL: NCT01730716
Title: A Phase II, Open-label, Dose Escalation and Safety Study of Human Spinal Cord Derived Neural Stem Cell Transplantation for the Treatment of Amyotrophic Lateral Sclerosis
Brief Title: Dose Escalation and Safety Study of Human Spinal Cord Derived Neural Stem Cell Transplantation for the Treatment of Amyotrophic Lateral Sclerosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neuralstem Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS2012-3
Record Dates: First submitted 2012-11-06; First posted 2012-11-21 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2013-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Human spinal cord derived neural stem cell transplantation; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgery (Experimental): There will be 5 sequential cohorts (Groups A-E) with 3 subjects in each cohort. Each cohort will follow a dose escalation plan. New patients will be enrolled into each group. No control group is included. All patients will received spinal cord injections of HSSC.
  Interventions: Device: Human spinal cord stem cell implantation

INTERVENTIONS:
Device: Human spinal cord stem cell implantation — Human spinal cord stem cell implantation in ALS patients.

SUMMARY:
The study is to determine the feasibility, safety, toxicity, and maximum tolerated (safe) dose of human spinal derived neural stem cell transplantation for the treatment of Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
These stem cells are called Human Spinal Stem Cells (HSSC) and have been engineered from the spinal cord of a single fetus electively aborted after 8 weeks of gestation. The tissue was obtained with the mother's consent. The cells will be transplanted into the ALS patient's spinal cord after laminectomy, an operation that removes bone surrounding the spine. After the spinal cord is exposed, a device manufactured for this purpose will be mounted onto the patient and will hold a syringe filled with the cells. The syringe will have a needle attached and the needle will enter the spinal cord at 5-10 locations injecting the cells. The device will minimize trauma to the spinal cord by the needle by making the puncture precise and steady and injecting the material at a slow and steady speed.

ALS is a universally fatal neurodegenerative condition that causes weakness leading to paralysis and death. Life expectancy is 2-5 years. The cause is unknown and there is no effective treatment. Previous research has shown that on autopsy, ALS patients are found to have increased levels of the amino acid glutamate accumulated in the brain and spinal cord. This increase is thought to be caused by a decrease in the glutamate transporter which normally "cleans up" glutamate from the cells. HSSC are known to express amino acid transporters and it is hoped that this action will reduce the toxicity of accumulated glutamate and benefit ALS patients. There is a second hypothesized benefit of the HSSC and that is their ability to secrete neurotrophic support factors. Neurotrophic factors support the health of nerves.

There will be 5 sequential cohorts (Groups A - E) with 3 subjects in each cohort. New patients will be enrolled into each group. No control group is included. All subjects will receive spinal cord injections of HSSC. All subjects will also be ambulatory with respiratory function greater than or equal to 50% supine and 60% seated of predicted normal and will receive bilateral injections at the C3 through C5 cervical segments. Subjects in Group E will receive bilateral injections at the L2 through L5 lumbar segments and then return approximately one-three months later to receive bilateral injections at the C3 through C5 cervical segments.

The dose escalation plan is as follows:

1. Group A: 3 ambulatory early-stage subjects with arm weakness but not paralysis, to receive bilateral C3 through C4 injections of 2x106 cells (10 injections x 2x105 cells/ injection)
2. Group B: 3 ambulatory early-stage subjects with arm weakness but not paralysis, to receive bilateral C3 through C5 injections of 4x106 cells (20 injections x 2x105 cells/ injection)
3. Group C: 3 ambulatory early-stage subjects with arm weakness but not paralysis, to receive bilateral C3 through C5 injections of 6x106 cells (20 injections x 3x105 cells/ injection)
4. Group D: 3 ambulatory early-stage subjects with arm weakness but not paralysis, to receive bilateral C3 through C5 injections of 8x106 cells (20 injections x 4x105 cells/ injection)
5. Group E: 3 ambulatory early-stage subjects with arm weakness but not paralysis, to receive bilateral L2 through L5 injections of 8x106 cells (20 injections of 4x105 cells/ injection) and then approximately 4-12 weeks later to receive bilateral C3 through C5 injections of 8x106 cells (20 injections of 4x105 cells/ injection.

Transition from one group to the next will be determined by review of available safety data by a Safety Monitoring Board (SMB) which will occur approximately one month post surgery of the last subject in the group. The study data will be collected for 6 months post stem cell transplantation of each study subject. However, all subjects will be followed clinically until death and all SAEs and post-study data will be collected and reported. Autopsy will be strongly encouraged for evaluation of pathology and presence of transplanted cells.

The treatment consists of laminectomy or laminoplasty of approximately two to three vertebral segments overlying either L2 through L4 (for Group E only) or C3 through C5 cord segments (for all Groups) in order to allow intraspinal injections of HSSC. Each injection will administer approximately 2, 3, or 4 x 105 cells in approximately 8.5 - 10 µL volume. The subjects will receive 5 or 10 injections at approximately 4 to 5mm intervals on each side of the cord, in total 10 or 20 injections. Each injection is completed in approximately 3 minutes. The total surgical time is expected to be approximately 3 to 5 hours. After the surgery, subjects will receive routine standard of care for laminectomy subjects who undergo an intradural procedure. Prior to and after the transplant, subjects will be required to remain on immunosuppressive therapy. Immunosuppressive therapy will consist of: 1) basiliximab (Simulect®) 20mg intravenously (IV) when the dura is opened, then again at day 4 post transplantation; 2) tacrolimus (Prograf®) initially dosed at a maximum of 0.1 mg/kg divided approximately every 12 hours by mouth (po) on post transplant day 1, and then maintained at a dose that provides a trough serum level of 4 to 8 ng/ml (adjusted for IV use as necessary); and 3) mycophenolate mofetil (CellCept®) started on post transplant day 1 at 500 mg approximately every 12 hours and progressively increased over 2 weeks to 1.0 gram by mouth (po) twice a day as tolerated. Dose escalation may be modified at the discretion of the site Principal Investigator (PI). Subjects will also receive an initial bolus dose of methylprednisolone 125 mg IV approximately 2 hours prior to the first injection. Beginning on post-operative day 1, the subject will receive oral prednisone 60 mg po daily (QD) for 7 days postoperatively, then progressively decreased over the next 21 days as follows: 40 mg/day for 7 days, 20 mg/day for 7 days, then 10 mg/day for 7 days. At 28 days, prednisone will be discontinued. All pre- and post-surgery immunosuppressive drugs will be administered as noted above, at the discretion of the site PI. If these subjects have previously discontinued mycophenolate mofetil and/or tacrolimus, they may be re-challenged as per the dosing described above, at the discretion of the site PI.

The decision to continue immunosuppression therapy will be at the discretion of the site PIs. Mycophenolate mofetil may be dosed down to half or discontinued prior to the end of the study period if the subject experiences adverse reactions to the immunosuppressive agents. If adverse reactions still persist, tacrolimus dose can be further reduced in half and then further considered to be discontinued. Any or all of the immunosuppressive agents may be reduced or stopped at the discretion of the site PI if it is suspected or determined that the immunosuppressive agent is the cause of toxicity and if symptoms of toxicity cannot be managed adequately with symptomatic treatment.

The study will proceed successively from Group A to Group E with a 4-week interval between Groups. The Safety Monitoring Board (SMB) will be convened at the end of the 4-week interval and review all available safety data. Based on the safety outcomes from the 3 subjects in each Group, the SMB will recommend, according to a predetermined rule, whether to enroll 3 new subjects into the next Group, to continue to collect additional information from the same Group, to enroll additional subjects into the same Group, or to suspend the study. Potential subjects will be recruited for the study but put on a waiting list until SMB approval of their treatment. The SMB will consist of 3 neurologists with expertise in ALS, 1 spinal neurosurgeon, 1 neurooncologist, 1 transplant immunologist, and the scientific director of the ALS Association.

Subjects will be assessed for adverse events including pain and infection, motor function, and quality of life. Additional assessments will be made to measure any postoperative changes from baseline in neurologic deficits, imaging studies, bladder or bowel function, allodynia, and neuropathic pain (see schedule of activities). Subjects will also undergo serial assessments of respiratory function (vital capacity (VC) and negative inspiratory force (NIF)), motor function (Ashworth Spasticity Scale, hand-held dynamometry and electrical impedance myography (EIM)), and respiratory function (diaphragm ultrasound). All subjects will undergo cardiac autonomic function testing at Day -14 to Day -2 pre-operatively, and at 1 and 3 months post-operatively to monitor for potential cardiac autonomic neuropathy.

There will be a lead-in period of at least 1 month period of clinical evaluations before surgery to estimate the slope of decline of clinical status. Measures during this lead-in time will be the ALSFRS-R, hand-held dynamometry/grip strength, Ashworth Spasticity Scale, VC and NIF, EIM, and diaphragm ultrasound.Subjects will be followed postoperatively at 2 and 4 weeks, and then at 3, 6, 9, 12, 15, 18, 21, and 24 months, and then at every 6 months thereafter until death.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to understand the requirements of the study, provide written informed consent, understand and provide written authorization for the use and disclosure of Protected Health Information (PHI) [per Health Insurance Portability and Accountability Act (HIPAA) Privacy Ruling] and comply with the study procedures.
2. Subjects with sporadic or familial ALS, meeting the definition of laboratory-supported probable, probable or definite ALS according to the World Federation of Neurology El Escorial Criteria (Appendix A). At the time of enrollment subjects should be within 24 months of symptom onset.
3. Age 18 years or older.
4. Females must have a negative serum pregnancy test and practice an acceptable method of contraception or be of non-childbearing potential (post-menopausal for at least 2 years or surgically sterile [hysterectomy, oophorectomy or surgical sterilization]).
5. Geographic accessibility to the study center and the ability to travel to the clinic for study visits.
6. Presence of a willing and able caregiver.
7. Medically able to undergo lumbar and/or cervical laminectomy or laminoplasty as determined by the site Principal Investigator and neurosurgeon.
8. Medically able to tolerate the immunosuppression regimen consisting of basiliximab, tacrolimus, mycophenolate mofetil, prednisone and methylprednisolone as determined by the site PI.
9. Agrees to the visit schedule as outlined in the informed consent.
10. Not taking riluzole (Rilutek®) or on a stable dose for ≥ 30 days.
11. Vital capacity ≥ 60% of predicted normal for age, height and gender measured in the seated position and ≥50% in supine position during the 7 days prior to surgery.
12. Ambulatory subjects with extremity weakness and/or spasticity due to ALS. Patients undergoing lumbar surgery must have demonstrable weakness or spasticity in one or both lower extremities. Patients undergoing cervical surgery must have demonstrable weakness or spasticity in one or both upper extremities, with at least antigravity strength. Subjects must have normal neck extensor and flexor strength.

Exclusion Criteria:

1. Etiology of paraplegia or weakness is due to causes other than ALS.
2. A positive result on the Panel Reactive Antibody (PRA) test, with the presence of specific HLA antibodies matching the HLA DNA profile of the donor cells.
3. Any known immunodeficiency syndrome.
4. Receipt of any investigational drug, device or biologic within 30 days of surgery.
5. Any concomitant medical disease or condition limiting the safety to participate:

   1. Coagulopathy
   2. Active uncontrolled infection
   3. Hypotension requiring vasopressor therapy
   4. Previous spinal surgery that the neurosurgeon deems to be an obstacle to the planned transplantation
   5. Skin breakdown over the site of surgery
   6. Malignancy (except for non-melanoma skin cancer)
   7. Spinal stenosis severe enough to preclude surgery (as determined by the neurosurgeon)
   8. Pre-existing kyphosis by preoperative MRI or X-ray
   9. Less than 5/5 grade in neck extension and strength test at the time of surgery.
6. Creatinine >1.5, liver function tests (SGOT/SGPT, Bilirubin, Alk Phos) > 2x upper limit of normal, hematocrit/hemoglobin < 30/10, total WBC < 4000, uncontrolled hypertension (systolic > 180 or diastolic > 100) or uncontrolled diabetes (defined as hemoglobin A1C >8), evidence of GI bleeding by hemoccult test, tuberculosis (TB test: PPD), serologic evidence of current infection with a hepatitis virus or human immunodeficiency virus (HIV).
7. Presence of any of the following conditions:

   1. Current drug abuse or alcoholism
   2. Unstable medical conditions
   3. Unstable psychiatric illness including psychosis and untreated major depression within 90 days of screening
8. Any condition or ALS disease phenotype that the site PI feels may interfere with participation in the study or in the interpretation of study endpoints.
9. Any condition that the neurosurgeon feels may pose complications for the surgery.
10. Known hypersensitivity to basiliximab, tacrolimus, mycophenolate mofetil, prednisone or methylprednisolone.
11. Inability to provide informed consent as determined by the site PI.
12. Inadequate family or caregiver support as determined by the site PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-12 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
To determine the safety of the maximum tolerated dose of human spinal cord-derived neural stem cell transplantation for the treatment of amyotrophic lateral sclerosis (ALS) assessed by the number and severity of adverse events. | Patients will be followed postoperatively for 24 months.
  The primary objective of the study is to determine the feasibility, safety, toxicity, and maximum tolerated (safe) dose of human spinal cord-derived neural stem cell transplantation for the treatment of amyotrophic lateral sclerosis (ALS).

SECONDARY OUTCOMES:
To evaluate neurologic deficits post spinal stem cell transplantation therapy. | Patients will be followed postoperatively for 24 months.
  The secondary objectives of the study are to evaluate spinal stem cell transplantation therapy in this patient population for: 1) attenuation of motor function loss; 2) maintenance of respiratory capacity; 3) stabilization of ALSFRS-R; 4) reduction of spasticity/rigidity if present; and 5) graft survival at autopsy if and when there is mortality.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan

REFERENCES:
- [Background] Glass JD, Boulis NM, Johe K, Rutkove SB, Federici T, Polak M, Kelly C, Feldman EL. Lumbar intraspinal injection of neural stem cells in patients with amyotrophic lateral sclerosis: results of a phase I trial in 12 patients. Stem Cells. 2012 Jun;30(6):1144-51. doi: 10.1002/stem.1079. PMID 22415942
- [Background] Riley J, Federici T, Polak M, Kelly C, Glass J, Raore B, Taub J, Kesner V, Feldman EL, Boulis NM. Intraspinal stem cell transplantation in amyotrophic lateral sclerosis: a phase I safety trial, technical note, and lumbar safety outcomes. Neurosurgery. 2012 Aug;71(2):405-16; discussion 416. doi: 10.1227/NEU.0b013e31825ca05f. PMID 22565043
- See also: Related Info — http://neuralstem.com